CLINICAL TRIAL: NCT00796653
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 48 Weeks of Once Daily Treatment of Orally Inhaled BI 1744 CL (5 µg [2 Actuations of 2.5 ug] and 10 ug [2 Actuations of 5 ug]) Delivered by the Respimat® Inhaler, and 48 Weeks of Twice Daily Foradil® (12 µg) Delivered by the Aerolizer® Inhaler, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Efficacy of BI 1744 CL in Patients With Chronic Obstructive Pulmonary Disease II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.14; 2008-001934-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Formoterol Fumarate

ARMS (4):
- Olodaterol (BI 1744) Low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Olodaterol (BI 1744) High (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Formoterol 12mcg (Active Comparator): 12mcg inhaled twice daily from the Aerolizer inhaler
  Interventions: Drug: Formoterol
- Placebo (Placebo Comparator): Olodaterol (BI 1744) placebo inhaled once daily from the Respimat inhaler and/or Formoterol placebo inhaled twice daily from the Aerolizer inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) Low
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) High
Drug: Formoterol — Active comparator with Olodaterol (BI 1744) on safety and efficacy in COPD patients
  Arms: Formoterol 12mcg
Drug: Placebo — Placebo devices for comparison with Olodaterol (BI 1744) on safety and efficacy in COPD patients
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the long-term efficacy and safety of once daily treatment of BI 1744 CL inhalation solution (5 and 10 mcg) delivered via the Respimat® inhaler, in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:post-bronchodilator FEV1<80% of predicted normal (ECSC) and a post-bronchodilator FEV1/FVC <70% at Visit 1
2. Male or female patients, 40 years of age or older
3. Patients must be current or ex-smokers with a smoking history of more than 10 pack years:

Exclusion criteria:

1. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT >x2 ULN, SGPT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN
2. Patients with a history of asthma and/or total blood eosinophil count greater than 600/mm3
3. Patients with thyrotoxicosis, paroxysmal tachycardia (>100 beats per minute)
4. Patients with a history of myocardial infarction within 1 year of screening visit, unstable or life-threatening cardiac arrhythmia, hospitalization for heart failure within the past year, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years, life-threatening pulmonary obstruction, cystic fibrosis, clinically evident bronchiectasis, significant alcohol or drug abuse
5. Patients who have undergone thoracotomy with pulmonary resection
6. Patients being treated with oral beta-adrenergics or oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
7. Patients who regularly use daytime oxygen therapy for more than one hour per day.
8. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
9. Pregnant or nursing women
10. Women of childbearing potential not using two effective methods of birth control (one barrier and one non-barrier).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 937 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (98):
- Argentina (5):
  - 1222.14.5004 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1222.14.5003 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1222.14.5001 Boehringer Ingelheim Investigational Site, Mendoza
  - 1222.14.5002 Boehringer Ingelheim Investigational Site, Quilmes
  - 1222.14.5005 Boehringer Ingelheim Investigational Site, San Juan Bautista
- Brazil (6):
  - 1222.14.5106 Boehringer Ingelheim Investigational Site, Florianópolis
  - 1222.14.5101 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1222.14.5103 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1222.14.5104 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1222.14.5102 Boehringer Ingelheim Investigational Site, Recife
  - 1222.14.5105 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (14):
  - 1222.14.4005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1222.14.4002 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 1222.14.4004 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1222.14.4009 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1222.14.4010 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1222.14.4008 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1222.14.4014 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1222.14.4007 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1222.14.4013 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1222.14.4001 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 1222.14.4012 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1222.14.4006 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1222.14.4015 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1222.14.4011 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Czechia (4):
  - 1222.14.6004 Boehringer Ingelheim Investigational Site, Brno
  - 1222.14.6003 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1222.14.6002 Boehringer Ingelheim Investigational Site, Kyjov
  - 1222.14.6001 Boehringer Ingelheim Investigational Site, Znojmo
- Denmark (3):
  - 1222.14.4602 Boehringer Ingelheim Investigational Site, Elsinore
  - 1222.14.4601 Boehringer Ingelheim Investigational Site, Hillerød
  - 1222.14.4603 Boehringer Ingelheim Investigational Site, Roskilde
- Finland (3):
  - 1222.14.4702 Boehringer Ingelheim Investigational Site, Espoo
  - 1222.14.4701 Boehringer Ingelheim Investigational Site, HUS
  - 1222.14.4703 Boehringer Ingelheim Investigational Site, Lohja
- Germany (12):
  - 1222.14.4106 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1222.14.4112 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.14.4103 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1222.14.4110 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1222.14.4108 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 1222.14.4107 Boehringer Ingelheim Investigational Site, Kelkheim
  - 1222.14.4114 Boehringer Ingelheim Investigational Site, Lübeck
  - 1222.14.4111 Boehringer Ingelheim Investigational Site, Mainz
  - 1222.14.4113 Boehringer Ingelheim Investigational Site, Minden
  - 1222.14.4109 Boehringer Ingelheim Investigational Site, Mönchengladbach
  - 1222.14.4104 Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - 1222.14.4105 Boehringer Ingelheim Investigational Site, Wiesloch
- 1222.14.5501 Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- India (11):
  - 1222.14.5412 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1222.14.5406 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1222.14.5402 Boehringer Ingelheim Investigational Site, Indore
  - 1222.14.5405 Boehringer Ingelheim Investigational Site, Jaipur
  - 1222.14.5409 Boehringer Ingelheim Investigational Site, Jaipur
  - 1222.14.5403 Boehringer Ingelheim Investigational Site, Mangalore
  - 1222.14.5407 Boehringer Ingelheim Investigational Site, Mysore
  - 1222.14.5404 Boehringer Ingelheim Investigational Site, Nagpur
  - 1222.14.5408 Boehringer Ingelheim Investigational Site, Noida
  - 1222.14.5401 Boehringer Ingelheim Investigational Site, Pune
  - 1222.14.5410 Boehringer Ingelheim Investigational Site, Vellore
- Italy (5):
  - 1222.14.4301 Boehringer Ingelheim Investigational Site, Cassano Delle Murge (ba)
  - 1222.14.4302 Boehringer Ingelheim Investigational Site, Genova
  - 1222.14.4304 Boehringer Ingelheim Investigational Site, Milan
  - 1222.14.4305 Boehringer Ingelheim Investigational Site, Parma
  - 1222.14.4303 Boehringer Ingelheim Investigational Site, Roma
- Malaysia (3):
  - 1222.14.5701 Boehringer Ingelheim Investigational Site, Georgetown, Pulau Pinang
  - 1222.14.5703 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1222.14.5702 Boehringer Ingelheim Investigational Site, Kuching, Sarawak
- Norway (2):
  - 1222.14.4802 Boehringer Ingelheim Investigational Site, Fredrikstad
  - 1222.14.4801 Boehringer Ingelheim Investigational Site, Ski
- Philippines (3):
  - 1222.14.5802 Boehringer Ingelheim Investigational Site, Iloilo City
  - 1222.14.5803 Boehringer Ingelheim Investigational Site, Iloilo City
  - 1222.14.5801 Boehringer Ingelheim Investigational Site, Manila
- Romania (3):
  - 1222.14.6103 Boehringer Ingelheim Investigational Site, Brasov
  - 1222.14.6102 Boehringer Ingelheim Investigational Site, Constanța
  - 1222.14.6101 Boehringer Ingelheim Investigational Site, Iași
- Russia (3):
  - 1222.14.6203 Boehringer Ingelheim Investigational Site, Petrozavodsk
  - 1222.14.6201 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1222.14.6202 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Africa (2):
  - 1222.14.4901 Boehringer Ingelheim Investigational Site, Cape Town
  - 1222.14.4902 Boehringer Ingelheim Investigational Site, Cape Town
- South Korea (6):
  - 1222.14.5301 Boehringer Ingelheim Investigational Site, Bucheon-si
  - 1222.14.5302 Boehringer Ingelheim Investigational Site, Seoul
  - 1222.14.5305 Boehringer Ingelheim Investigational Site, Seoul
  - 1222.14.5306 Boehringer Ingelheim Investigational Site, Seoul
  - 1222.14.5304 Boehringer Ingelheim Investigational Site, Uijeongbu-si
  - 1222.14.5303 Boehringer Ingelheim Investigational Site, Wŏnju
- Spain (6):
  - 1222.14.4401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1222.14.4402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1222.14.4406 Boehringer Ingelheim Investigational Site, Madrid
  - 1222.14.4405 Boehringer Ingelheim Investigational Site, Mérida
  - 1222.14.4403 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1222.14.4407 Boehringer Ingelheim Investigational Site, Terrassa (Barcelona)
- Sweden (3):
  - 1222.14.4501 Boehringer Ingelheim Investigational Site, Boden
  - 1222.14.4503 Boehringer Ingelheim Investigational Site, Göteboerg
  - 1222.14.4502 Boehringer Ingelheim Investigational Site, Lund
- Thailand (3):
  - 1222.14.5904 Boehringer Ingelheim Investigational Site, Bangkok
  - 1222.14.5901 Boehringer Ingelheim Investigational Site, Khon Kaen
  - 1222.14.5902 Boehringer Ingelheim Investigational Site, Songkhla

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Andreas S, Bothner U, de la Hoz A, Kloer I, Trampisch M, Alter P. A Post Hoc Holter ECG Analysis of Olodaterol and Formoterol in Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1955-1965. doi: 10.2147/COPD.S246353. eCollection 2020. PMID 32848381
- [Derived] Andreas S, Bothner U, Trampisch M, Haensel M, Buhl R, Alter P. Effect of long-acting beta2-agonists olodaterol and formoterol on heart rate and blood pressure in chronic obstructive pulmonary disease patients. Pulm Pharmacol Ther. 2018 Oct;52:1-6. doi: 10.1016/j.pupt.2018.08.002. Epub 2018 Aug 2. PMID 30077810
- [Derived] Koch A, Pizzichini E, Hamilton A, Hart L, Korducki L, De Salvo MC, Paggiaro P. Lung function efficacy and symptomatic benefit of olodaterol once daily delivered via Respimat(R) versus placebo and formoterol twice daily in patients with GOLD 2-4 COPD: results from two replicate 48-week studies. Int J Chron Obstruct Pulmon Dis. 2014 Jul 5;9:697-714. doi: 10.2147/COPD.S62502. eCollection 2014. PMID 25045258

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were randomized but not treated due to withdrawn consent and findings on pre-dose ECG prior to receiving study medication.
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olodaterol (Olo) 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olodaterol (Olo) 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Form 12 mcg: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Period: Overall Study
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Form 12 mcg
Started | 235 | 232 | 234 | 233
Completed | 184 | 195 | 198 | 193
Not Completed | 51 | 37 | 36 | 40
Not completed — Adverse Event | 19 | 16 | 16 | 16
Not completed — Lost to Follow-up | 2 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 16 | 8 | 8 | 13
Not completed — Lack of Efficacy | 8 | 1 | 3 | 2
Not completed — Non compliance with protocol | 2 | 2 | 0 | 2
Not completed — Other reason not described above | 4 | 9 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Total: Total of all reporting groups
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg | Total
Number analyzed (Participants) | 235 | 232 | 234 | 233 | 934
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.8) | 63.7 (8.8) | 63.8 (8.5) | 65.0 (8.2) | 64.183 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 45 | 50 | 41 | 176
  Male | 195 | 187 | 184 | 192 | 758
Tiotropium (Tio) Use Stratum [Number; unit: Number of participants]
  Non-tiotropium | 173 | 174 | 172 | 174 | 693
  Tiotropium | 62 | 58 | 62 | 59 | 241

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 24 Weeks
Description: Response was defined as change from baseline. Baseline FEV1 was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first am dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 24
Population: Full analysis set (FAS). FAS is defined as all randomized patients who received at least one dose of treatment and had both baseline data and at least one post-baseline measurement at or before 24 weeks for any of the co-primary efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | -0.013 (0.014) | 0.116 (0.014) | 0.140 (0.014) | 0.137 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects,baseline, baseline-by-visit as fixed covariates, patient as random effect; Mean Difference (Final Values) = 0.129, 95% CI [0.091 to 0.167], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.154, 95% CI [0.116 to 0.191], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI [0.112 to 0.188], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

2. Primary Outcome: Trough FEV1 Response at Week 24
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FEV1s if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 24.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.055 (0.014) | -0.003 (0.014) | 0.014 (0.014) | -0.013 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.053, 95% CI [0.015 to 0.090], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI [0.032 to 0.106], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0270, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.042, 95% CI [0.005 to 0.080], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

3. Primary Outcome: Mahler Transitional Dyspnea Index Focal Score at 24 Weeks
Description: Mahler Transitional Dyspnea Index (TDI) focal score measures 3 components of dyspnea that evoke dyspnea in daily living: Functional Impairment, Magnitude of Task, and Magnitude of Effort. The TDI measures the change from the baseline assessment ranging from -9 (most deterioration) to +9 (most improvement).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 1.102 (0.229) | 1.504 (0.225) | 1.521 (0.225) | 1.703 (0.228)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1999, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.402, 95% CI [-0.213 to 1.018], Standard Error of Mean 0.314 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1818, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.419, 95% CI [-0.196 to 1.035], Standard Error of Mean 0.314 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0572, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.602, 95% CI [-0.019 to 1.222], Standard Error of Mean 0.316 — Form 12 mcg minus Placebo

4. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 24 Weeks
Description: Saint George's Respiratory Questionnaire (SGRQ) measures the impact of COPD on overall health, daily life, and perceived well-being ranging from 0 (no limitations) to 100 (most limitations).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 202 | 216 | 212 | 206
score on a scale | 42.120 (0.995) | 38.970 (0.965) | 38.597 (0.969) | 40.704 (0.984)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0197, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.150, 95% CI [-5.796 to -0.503], Standard Error of Mean 1.349 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0094, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.524, 95% CI [-6.180 to -0.867], Standard Error of Mean 1.354 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2995, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.416, 95% CI [-4.093 to 1.261], Standard Error of Mean 1.365 — Form 12 mcg minus Placebo

5. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 48 Weeks
Description: as for outcome 4
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 202 | 216 | 212 | 206
score on a scale | 39.914 (1.022) | 39.562 (0.986) | 38.824 (0.991) | 40.025 (0.996)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.7995, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.352, 95% CI [-3.068 to 2.365], Standard Error of Mean 1.385 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.4336, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.090, 95% CI [-3.818 to 1.639], Standard Error of Mean 1.391 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.9365, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.111, 95% CI [-2.625 to 2.848], Standard Error of Mean 1.395 — Form 12 mcg minus Placebo

6. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 12 Weeks
Description: as for outcome 4
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 202 | 216 | 212 | 206
score on a scale | 42.679 (0.983) | 40.054 (0.955) | 40.190 (0.963) | 39.521 (0.975)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0491, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.625, 95% CI [-5.241 to -0.010], Standard Error of Mean 1.333 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0636, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.489, 95% CI [-5.119 to 0.141], Standard Error of Mean 1.341 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0194, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.158, 95% CI [-5.806 to -0.511], Standard Error of Mean 1.350 — Form 12 mcg minus Placebo

7. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 24 Weeks for Combined Analysis
Description: Saint George's Respiratory Questionnaire (SGRQ) measures the impact of COPD on overall health, daily life, and perceived well-being ranging from 0 (no limitations) to 100 (most limitations). This is a combined analysis of the data from NCT00793624 and NCT00796653 showing adjusted values using a MMRM model.
Time Frame: Baseline, Week 24
Population: Full analysis sets (FAS) of the trials NCT00793624 and NCT00796653. FAS is defined as all randomized patients who received at least one dose of treatment and had both baseline data and at least one post-baseline measurement at or before 24 weeks for any of the co-primary efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 387 | 416 | 414 | 408
score on a scale | 41.639 (0.718) | 38.794 (0.693) | 38.205 (0.695) | 40.391 (0.699)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Olo 5 mcg minus placebo; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.846, 95% CI 2-sided [-4.751 to -0.940], Standard Error of Mean 0.972
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Olo 10 mcg minus placebo; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.434, 95% CI 2-sided [-5.343 to -1.525], Standard Error of Mean 0.973
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Form 12 mcg minus placebo; Test type: Superiority or Other; p = 0.2009, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.248, 95% CI 2-sided [-3.161 to 0.665], Standard Error of Mean 0.976

8. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 2 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.021 (0.013) | 0.181 (0.014) | 0.214 (0.013) | 0.183 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.160, 95% CI [0.123 to 0.196], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.193, 95% CI [0.157 to 0.229], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.162, 95% CI [0.126 to 0.199], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

9. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 6 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | -0.010 (0.014) | 0.162 (0.014) | 0.181 (0.014) | 0.174 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.136 to 0.209], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.155 to 0.228], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.184, 95% CI [0.148 to 0.221], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

10. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 12 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | -0.008 (0.014) | 0.138 (0.014) | 0.167 (0.014) | 0.163 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.145, 95% CI [0.108 to 0.182], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.175, 95% CI [0.138 to 0.212], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.170, 95% CI [0.133 to 0.208], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

11. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 48 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | -0.025 (0.014) | 0.093 (0.014) | 0.116 (0.014) | 0.104 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.118, 95% CI [0.080 to 0.156], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.103 to 0.180], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.129, 95% CI [0.091 to 0.168], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

12. Secondary Outcome: Trough FEV1 Response at Week 2
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 2.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.016 (0.013) | 0.053 (0.013) | 0.103 (0.013) | 0.033 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI [0.033 to 0.105], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.119, 95% CI [0.083 to 0.155], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.049, 95% CI [0.013 to 0.085], Standard Error of Mean 0.018 — Form 12 mcg minus Placebo

13. Secondary Outcome: Trough FEV1 Response at Week 6
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 6.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.036 (0.013) | 0.047 (0.013) | 0.068 (0.013) | 0.034 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.084, 95% CI [0.048 to 0.120], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.104, 95% CI [0.068 to 0.141], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.070, 95% CI [0.034 to 0.106], Standard Error of Mean 0.018 — Form 12 mcg minus Placebo

14. Secondary Outcome: Trough FEV1 Response at Week 12
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 12.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.041 (0.014) | 0.018 (0.013) | 0.052 (0.013) | 0.024 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [0.022 to 0.095], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.093, 95% CI [0.057 to 0.130], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.065, 95% CI [0.028 to 0.101], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

15. Secondary Outcome: Trough FEV1 Response at Week 18
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 18.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.036 (0.014) | 0.013 (0.014) | 0.049 (0.013) | 0.015 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.050, 95% CI [0.013 to 0.087], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.086, 95% CI [0.049 to 0.122], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.051, 95% CI [0.014 to 0.088], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

16. Secondary Outcome: Trough FEV1 Response at Week 32
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 32.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.039 (0.014) | 0.023 (0.014) | 0.034 (0.014) | 0.009 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.062, 95% CI [0.025 to 0.100], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.073, 95% CI [0.035 to 0.110], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0117, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.048, 95% CI [0.011 to 0.086], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

17. Secondary Outcome: Trough FEV1 Response at Week 40
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 40.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.043 (0.014) | 0.019 (0.014) | 0.041 (0.014) | 0.013 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.062, 95% CI [0.024 to 0.099], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.084, 95% CI [0.047 to 0.122], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.056, 95% CI [0.019 to 0.094], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

18. Secondary Outcome: Trough FEV1 Response at Week 48
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 48.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.060 (0.014) | -0.016 (0.014) | -0.001 (0.014) | -0.024 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.044, 95% CI [0.006 to 0.082], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [0.021 to 0.097], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0664, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.036, 95% CI [-0.002 to 0.074], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

19. Secondary Outcome: Peak FEV1 (0-3h) Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.099 (0.014) | 0.260 (0.014) | 0.278 (0.014) | 0.253 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.122 to 0.199], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.178, 95% CI [0.140 to 0.216], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.153, 95% CI [0.115 to 0.191], Standard Error of Mean 0.019 — Form 12 mcg minus Placebo

20. Secondary Outcome: Peak FEV1 (0-3h) Response After 6 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.066 (0.014) | 0.235 (0.014) | 0.248 (0.014) | 0.242 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.168, 95% CI [0.130 to 0.207], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.181, 95% CI [0.143 to 0.220], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.176, 95% CI [0.137 to 0.214], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

21. Secondary Outcome: Peak FEV1 (0-3h) Response After 12 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.064 (0.014) | 0.206 (0.014) | 0.232 (0.014) | 0.228 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.103 to 0.180], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.168, 95% CI [0.129 to 0.207], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.125 to 0.203], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

22. Secondary Outcome: Peak FEV1 (0-3h) Response After 24 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.060 (0.015) | 0.183 (0.014) | 0.211 (0.014) | 0.203 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.123, 95% CI [0.084 to 0.163], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.151, 95% CI [0.112 to 0.191], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.143, 95% CI [0.104 to 0.183], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

23. Secondary Outcome: Peak FEV1 (0-3h) Response After 48 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.052 (0.015) | 0.163 (0.015) | 0.178 (0.015) | 0.170 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.112, 95% CI [0.071 to 0.152], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.126, 95% CI [0.086 to 0.166], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.118, 95% CI [0.078 to 0.158], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

24. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 2 Weeks
Description: Response was defined as change from baseline. Baseline FVC was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first am dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FVC AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.082 (0.025) | 0.312 (0.025) | 0.332 (0.025) | 0.348 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.231, 95% CI [0.162 to 0.299], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.250, 95% CI [0.182 to 0.318], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.266, 95% CI [0.198 to 0.334], Standard Error of Mean 0.035 — Form 12 mcg minus Placebo

25. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 6 Weeks
Description: as for outcome 24
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.027 (0.025) | 0.277 (0.026) | 0.276 (0.025) | 0.307 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.251, 95% CI [0.182 to 0.320], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.249, 95% CI [0.180 to 0.318], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.281, 95% CI [0.212 to 0.350], Standard Error of Mean 0.035 — Form 12 mcg minus Placebo

26. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 12 Weeks
Description: as for outcome 24
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.006 (0.026) | 0.235 (0.026) | 0.253 (0.026) | 0.280 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.229, 95% CI [0.159 to 0.299], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.247, 95% CI [0.177 to 0.317], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.275, 95% CI [0.205 to 0.345], Standard Error of Mean 0.036 — Form 12 mcg minus Placebo

27. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 24 Weeks
Description: as for outcome 24
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.012 (0.026) | 0.212 (0.026) | 0.225 (0.026) | 0.253 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.199, 95% CI [0.128 to 0.270], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.213, 95% CI [0.142 to 0.283], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.241, 95% CI [0.170 to 0.312], Standard Error of Mean 0.036 — Form 12 mcg minus Placebo

28. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 48 Weeks
Description: as for outcome 24
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | -0.036 (0.027) | 0.182 (0.026) | 0.201 (0.026) | 0.184 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.218, 95% CI [0.146 to 0.290], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.237, 95% CI [0.166 to 0.309], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.220, 95% CI [0.148 to 0.292], Standard Error of Mean 0.037 — Form 12 mcg minus Placebo

29. Secondary Outcome: Trough FVC Response at Week 2
Description: Response was defined as change from baseline. Baseline trough FVC was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FVC is defined as the FVC performed at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FVCs if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | 0.030 (0.026) | 0.118 (0.026) | 0.173 (0.026) | 0.111 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0133, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.088, 95% CI [0.018 to 0.157], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.143, 95% CI [0.073 to 0.212], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0212, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI [0.012 to 0.151], Standard Error of Mean 0.035 — Form 12 mcg minus Placebo

30. Secondary Outcome: Trough FVC Response at Week 6
Description: as for outcome 29
Time Frame: as for outcome 13
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.014 (0.026) | 0.113 (0.026) | 0.101 (0.026) | 0.085 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.127, 95% CI [0.057 to 0.197], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI [0.045 to 0.185], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.099, 95% CI [0.029 to 0.169], Standard Error of Mean 0.036 — Form 12 mcg minus Placebo

31. Secondary Outcome: Trough FVC Response at Week 12
Description: as for outcome 29
Time Frame: as for outcome 14
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.041 (0.026) | 0.062 (0.026) | 0.062 (0.026) | 0.070 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.032 to 0.173], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0046, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.102, 95% CI [0.032 to 0.173], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.110, 95% CI [0.039 to 0.181], Standard Error of Mean 0.036 — Form 12 mcg minus Placebo

32. Secondary Outcome: Trough FVC Response at Week 18
Description: as for outcome 29
Time Frame: as for outcome 15
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.014 (0.027) | 0.084 (0.026) | 0.107 (0.026) | 0.064 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [0.026 to 0.169], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.121, 95% CI [0.050 to 0.193], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0339, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.078, 95% CI [0.006 to 0.149], Standard Error of Mean 0.037 — Form 12 mcg minus Placebo

33. Secondary Outcome: Trough FVC Response at Week 24
Description: as for outcome 29
Time Frame: as for outcome 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.044 (0.027) | 0.023 (0.026) | 0.019 (0.026) | -0.005 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0718, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.066, 95% CI [-0.006 to 0.139], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0863, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.063, 95% CI [-0.009 to 0.135], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2982, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.038, 95% CI [-0.034 to 0.111], Standard Error of Mean 0.037 — Form 12 mcg minus Placebo

34. Secondary Outcome: Trough FVC Response at Week 32
Description: as for outcome 29
Time Frame: as for outcome 16
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.007 (0.027) | 0.081 (0.027) | 0.063 (0.027) | 0.036 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0190, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.087, 95% CI [0.014 to 0.160], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0601, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.070, 95% CI [-0.003 to 0.143], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2573, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.042, 95% CI [-0.031 to 0.115], Standard Error of Mean 0.037 — Form 12 mcg minus Placebo

35. Secondary Outcome: Trough FVC Response at Week 40
Description: as for outcome 29
Time Frame: as for outcome 17
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.016 (0.027) | 0.071 (0.027) | 0.105 (0.027) | 0.037 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0200, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.087, 95% CI [0.014 to 0.160], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.121, 95% CI [0.047 to 0.194], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.1598, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.053, 95% CI [-0.021 to 0.126], Standard Error of Mean 0.037 — Form 12 mcg minus Placebo

36. Secondary Outcome: Trough FVC Response at Week 48
Description: as for outcome 29
Time Frame: as for outcome 18
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 232 | 229 | 228 | 229
Liter | -0.069 (0.027) | 0.012 (0.027) | 0.032 (0.027) | -0.031 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0307, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.081, 95% CI [0.008 to 0.155], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.101, 95% CI [0.027 to 0.175], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.3147, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.038, 95% CI [-0.036 to 0.112], Standard Error of Mean 0.038 — Form 12 mcg minus Placebo

37. Secondary Outcome: Peak FVC (0-3h) Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline peak FVC was defined as the mean of the available pre-dose peak FVC values prior to first dose of randomized treatment. Peak FVC (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 19
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.247 (0.027) | 0.480 (0.027) | 0.476 (0.027) | 0.495 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.233, 95% CI [0.160 to 0.306], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.229, 95% CI [0.156 to 0.302], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.248, 95% CI [0.175 to 0.321], Standard Error of Mean 0.037 — Form 12 mcg minus Placebo

38. Secondary Outcome: Peak FVC (0-3h) Response After 6 Weeks
Description: as for outcome 37
Time Frame: as for outcome 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.196 (0.027) | 0.443 (0.027) | 0.417 (0.027) | 0.450 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.247, 95% CI [0.174 to 0.321], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.221, 95% CI [0.148 to 0.295], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.254, 95% CI [0.180 to 0.328], Standard Error of Mean 0.038 — Form 12 mcg minus Placebo

39. Secondary Outcome: Peak FVC (0-3h) Response After 12 Weeks
Description: as for outcome 37
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.171 (0.028) | 0.386 (0.027) | 0.396 (0.027) | 0.436 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.215, 95% CI [0.141 to 0.289], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.226, 95% CI [0.151 to 0.300], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.265, 95% CI [0.191 to 0.340], Standard Error of Mean 0.038 — Form 12 mcg minus Placebo

40. Secondary Outcome: Peak FVC (0-3h) Response After 24 Weeks
Description: as for outcome 37
Time Frame: as for outcome 22
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.189 (0.028) | 0.371 (0.028) | 0.369 (0.028) | 0.397 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.182, 95% CI [0.106 to 0.258], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.180, 95% CI [0.105 to 0.256], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.207, 95% CI [0.132 to 0.283], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

41. Secondary Outcome: Peak FVC (0-3h) Response After 48 Weeks
Description: as for outcome 37
Time Frame: as for outcome 23
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
Liter | 0.137 (0.029) | 0.325 (0.028) | 0.352 (0.028) | 0.329 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.188, 95% CI [0.111 to 0.265], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.214, 95% CI [0.138 to 0.291], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.115 to 0.269], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

42. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) at Week 24
Description: Weekly mean pre-dose morning and evening PEFR. Results are from non-MMRM ANCOVA models by week, with Last observation carried forward (LOCF) up to each week. Fixed effects include treatment, tiotropium, strata and baseline.
Time Frame: Week 24
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 233 | 230 | 233 | 232
L/min
  morning PEFR (N=225, 227, 226, 224) | 196.789 (3.270) | 210.496 (3.253) | 217.660 (3.274) | 211.038 (3.299)
  evening PEFR (N=224, 223, 227, 222) | 202.505 (3.281) | 219.905 (3.289) | 225.380 (3.281) | 218.321 (3.321)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.0021, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 13.707, 95% CI 2-sided [5.004 to 22.411], Standard Error of Mean 4.435
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 20.871, 95% CI 2-sided [12.158 to 29.584], Standard Error of Mean 4.440
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.0014, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 14.249, 95% CI 2-sided [5.506 to 22.991], Standard Error of Mean 4.454
Statistical Analysis 4: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 17.400, 95% CI 2-sided [8.640 to 26.160], Standard Error of Mean 4.463
Statistical Analysis 5: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 22.875, 95% CI 2-sided [14.153 to 31.596], Standard Error of Mean 4.444
Statistical Analysis 6: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0004, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 15.816, 95% CI 2-sided [7.032 to 24.599], Standard Error of Mean 4.475

43. Secondary Outcome: Use of Rescue Medication at Week 24
Description: Mean number of puffs of rescue medication used per day (daytime/nighttime/total)
Time Frame: Week 24
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 227 | 228 | 229 | 224
Number of puffs
  Daytime | 1.189 (0.089) | 1.036 (0.089) | 0.923 (0.089) | 0.967 (0.090)
  Nighttime | 1.713 (0.112) | 1.435 (0.111) | 1.348 (0.112) | 1.393 (0.113)
  Total | 2.893 (0.187) | 2.470 (0.187) | 2.277 (0.188) | 2.353 (0.190)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.2057, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.153, 95% CI 2-sided [-0.391 to -0.084], Standard Error of Mean 0.121
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.0284, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.266, 95% CI 2-sided [-0.504 to -0.028], Standard Error of Mean 0.121
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.0685, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.222, 95% CI 2-sided [-0.461 to 0.017], Standard Error of Mean 0.122
Statistical Analysis 4: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0674, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.278, 95% CI 2-sided [-0.576 to 0.020], Standard Error of Mean 0.152
Statistical Analysis 5: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0163, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.365, 95% CI 2-sided [-0.662 to -0.067], Standard Error of Mean 0.0163
Statistical Analysis 6: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0364, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.320, 95% CI 2-sided [-0.620 to -0.020], Standard Error of Mean 0.153
Statistical Analysis 7: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean daily (24h) rescue use; Test type: Superiority or Other; p = 0.0959, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.424, 95% CI 2-sided [-0.922 to 0.075], Standard Error of Mean 0.254
Statistical Analysis 8: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean daily (24h) rescue use; Test type: Superiority or Other; p = 0.0155, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.616, 95% CI 2-sided [-1.115 to -0.117], Standard Error of Mean 0.254
Statistical Analysis 9: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean daily (24h) rescue use; Test type: Superiority or Other; p = 0.0347, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.541, 95% CI 2-sided [-1.042 to -0.039], Standard Error of Mean 0.256

44. Secondary Outcome: Patient's Global Rating (PGR) at 6 Weeks
Description: Patient's Global Rating (PGR) was a patient assessment of their health (respiratory condition) at each visit (compared to the day before they started study drug) and ranged from 1 (very much better) to 7 (very much worse).
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 224 | 225 | 225 | 221
score on a scale | 3.4 (0.1) | 3.1 (0.1) | 3.2 (0.1) | 3.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0164, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.0], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0196, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.0], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

45. Secondary Outcome: Patient's Global Rating (PGR) at 12 Weeks
Description: as for outcome 44
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 224 | 225 | 225 | 221
score on a scale | 3.3 (0.1) | 3.1 (0.1) | 3.0 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0388, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.0], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0053, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

46. Secondary Outcome: Patient's Global Rating (PGR) at 24 Weeks
Description: as for outcome 44
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 224 | 225 | 225 | 221
score on a scale | 3.3 (0.1) | 3.1 (0.1) | 3.1 (0.1) | 3.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0555, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0122, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0144, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.1], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

47. Secondary Outcome: Patient's Global Rating (PGR) at 48 Weeks
Description: as for outcome 44
Time Frame: Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 224 | 225 | 225 | 221
score on a scale | 3.2 (0.1) | 3.2 (0.1) | 3.0 (0.1) | 3.2 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.5707, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.1, 95% CI [-0.3 to 0.1], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0814, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.7413, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.0, 95% CI [-0.2 to 0.2], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

48. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 6 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 0.980 (0.221) | 1.417 (0.221) | 1.686 (0.222) | 1.444 (0.224)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1524, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.437, 95% CI [-0.162 to 1.036], Standard Error of Mean 0.305 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0211, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.706, 95% CI [0.106 to 1.307], Standard Error of Mean 0.306 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.1314, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.464, 95% CI [-0.139 to 1.066], Standard Error of Mean 0.307 — Form 12 mcg minus Placebo

49. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 12 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 1.080 (0.224) | 1.742 (0.222) | 1.747 (0.224) | 1.499 (0.226)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0319, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.662, 95% CI [0.057 to 1.267], Standard Error of Mean 0.308 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0312, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.667, 95% CI [0.060 to 1.274], Standard Error of Mean 0.310 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.1777, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.419, 95% CI [-0.191 to 1.029], Standard Error of Mean 0.311 — Form 12 mcg minus Placebo

50. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 18 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 1.0454 (0.227) | 1.470 (0.223) | 1.537 (0.224) | 1.579 (0.227)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1714, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.425, 95% CI [-0.184 to 1.035], Standard Error of Mean 0.311 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1142, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.492, 95% CI [-0.119 to 1.103], Standard Error of Mean 0.312 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0888, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.534, 95% CI [-0.081 to 1.150], Standard Error of Mean 0.314 — Form 12 mcg minus Placebo

51. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 32 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 1.168 (0.232) | 1.658 (0.228) | 1.522 (0.228) | 1.477 (0.229)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1235, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.490, 95% CI [-0.134 to 1.113], Standard Error of Mean 0.318 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2666, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.354, 95% CI [-0.271 to 0.978], Standard Error of Mean 0.318 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.3335, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.309, 95% CI [-0.317 to 0.934], Standard Error of Mean 0.319 — Form 12 mcg minus Placebo

52. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 40 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 1.064 (0.234) | 1.377 (0.229) | 1.545 (0.229) | 1.178 (0.231)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3287, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.313, 95% CI [-0.315 to 0.941], Standard Error of Mean 0.320 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1341, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.481, 95% CI [-0.148 to 1.109], Standard Error of Mean 0.321 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.7220, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.114, 95% CI [-0.516 to 0.745], Standard Error of Mean 0.322 — Form 12 mcg minus Placebo

53. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 48 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 221 | 221 | 220 | 215
score on a scale | 1.113 (0.234) | 1.510 (0.231) | 1.831 (0.230) | 1.280 (0.232)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2176, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.397, 95% CI [-0.234 to 1.027], Standard Error of Mean 0.322 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0258, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.718, 95% CI [0.087 to 1.348], Standard Error of Mean 0.323 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.6044, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.167, 95% CI [-0.466 to 0.800], Standard Error of Mean 0.323 — Form 12 mcg minus Placebo

54. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.
Time Frame: Baseline to end of study at 48 weeks.
Measure: Mean (95% Confidence Interval); unit: Days
Groups:
- Placebo (Tiotropium): Matching Placebo delivered by the Respimat Inhaler - tiotropium use stratum
- Placebo (Non-tiotropium): Matching Placebo delivered by the Respimat Inhaler - non-tiotropium use stratum.
- Olo 5 mcg qd (Tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 5 mcg qd (Non-tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
- Olo 10 mcg qd (Tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 10 mcg qd(Non-tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
- Form 12 mcg (Tiotropium): Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler - tiotropium stratum
- Form 12 mcg (Non-tiotropium): Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler - non-tiotropium stratum
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium) | Form 12 mcg (Tiotropium) | Form 12 mcg (Non-tiotropium)
Number analyzed (Participants) | 61 | 174 | 59 | 173 | 59 | 175 | 58 | 175
Days | 173 [74.0 to 298.0] | 177 [118.0 to 221.0] | 252 [164.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 270 [180.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 252 [92.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 234 [184.0 to 326.0] | 149 [106.0 to 217.0] | 232 [161.0 to 368.0]
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Olo 5 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.1946, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.802, 95% CI [0.580 to 1.111], Standard Error of Mean 0.133 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Olo 10 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.4071, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.872, 95% CI [0.634 to 1.198], Standard Error of Mean 0.141 — Comparison of Olo 10 mcg qd to placebo across stratum
Statistical Analysis 3: Comparison: Placebo (Tiotropium) vs Form 12 mcg (Tiotropium); Test type: Superiority or Other; p = 0.6404, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.922, 95% CI [0.670 to 1.267], Standard Error of Mean 0.150 — Comparison of Form 12 mcg to placebo across stratum

55. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (CPOD) Exacerbation Leading to Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.
Time Frame: Baseline to end of study at 48 weeks.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium) | Form 12 mcg (Tiotropium) | Form 12 mcg (Non-tiotropium)
Number analyzed (Participants) | 61 | 174 | 59 | 173 | 59 | 175 | 58 | 175
Days | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 368.0 [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Olo 5 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.2942, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.685, 95% CI [0.336 to 1.399], Standard Error of Mean 0.249 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Olo 10 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.8594, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.947, 95% CI [0.493 to 1.820], Standard Error of Mean 0.316 — Comparison of Olo 10 mcg qd to placebo across stratum
Statistical Analysis 3: Comparison: Placebo (Tiotropium) vs Form 12 mcg (Tiotropium); Test type: Superiority or Other; p = 0.5466, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.803, 95% CI [0.405 to 1.593], Standard Error of Mean 0.281 — Comparison of Form 12 mcg to placebo across stratum

56. Secondary Outcome: Time to First Moderate Chronic Obstructive Pulmonary Disease (CPOD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.
Time Frame: Baseline to end of study at 48 weeks.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium) | Form 12 mcg (Tiotropium) | Form 12 mcg (Non-tiotropium)
Number analyzed (Participants) | 61 | 174 | 59 | 173 | 59 | 175 | 58 | 175
Days | 176 [75.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 214 [144.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 264 [164.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 312 [205.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 324 [126.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 327 [237.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 190 [112.0 to 260.0] | 325 [181.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Olo 5 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.2494, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.807, 95% CI [0.566 to 1.150], Standard Error of Mean 0.146 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Olo 10 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.2006, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.791, 95% CI [0.555 to 1.126], Standard Error of Mean 0.143 — Comparison of Olo 10 mcg qd to placebo across stratum
Statistical Analysis 3: Comparison: Placebo (Tiotropium) vs Form 12 mcg (Tiotropium); Test type: Superiority or Other; p = 0.5795, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.903, 95% CI [0.637 to 1.279], Standard Error of Mean 0.160 — Comparison of Form 12 mcg to placebo across stratum

57. Secondary Outcome: Number of COPD Exacerbations
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD ex. per patient year
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 235 | 232 | 234 | 233
Number of COPD ex. per patient year | 0.6890 (0.0829) | 0.5409 (0.0690) | 0.5947 (0.0736) | 0.7325 (0.0861)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1571, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.7850, 95% CI [0.5613 to 1.0979], Standard Error of Mean 0.1342 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.3814, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.8631, 95% CI [0.6205 to 1.2005], Standard Error of Mean 0.1451 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.7098, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.0631, 95% CI [0.7699 to 1.4680], Standard Error of Mean 0.1748 — Form 12 mcg minus Placebo

58. Secondary Outcome: Number of COPD Exacerbations Requiring Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD ex. per patient year
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 235 | 232 | 234 | 233
Number of COPD ex. per patient year | 0.0986 (0.0258) | 0.0781 (0.0221) | 0.0993 (0.0253) | 0.1025 (0.0262)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.5326, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.7925, 95% CI [0.3814 to 1.6464], Standard Error of Mean 0.2952 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.9824, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.0078, 95% CI [0.5038 to 2.0160], Standard Error of Mean 0.3560 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.9112, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.0403, 95% CI [0.5194 to 2.0832], Standard Error of Mean 0.3681 — Form 12 mcg minus Placebo

59. Secondary Outcome: Number of Moderate Chronic Obstructive Pulmonary Disease (CPOD) Exacerbations
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD ex. per patient year
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 235 | 232 | 234 | 233
Number of COPD ex. per patient year | 0.5548 (0.0719) | 0.4128 (0.0578) | 0.4351 (0.0601) | 0.5415 (0.0699)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1136, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.7440, 95% CI [0.5158 to 1.0733], Standard Error of Mean 0.1389 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1887, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.7842, 95% CI [0.5456 to 1.1271], Standard Error of Mean 0.1449 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.8925, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.9761, 95% CI [0.6869 to 1.3870], Standard Error of Mean 0.1747 — Form 12 mcg minus Placebo

60. Secondary Outcome: Changes in Safety Parameters Related to Treatment
Description: Occurence of cardiac disorders and investigations related to treatment.
Time Frame: 48 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 235 | 232 | 234 | 233
percentage of participants
  Atrial fibrillation | 0.9 | 0.0 | 0.9 | 0.0
  Sinus tachycardia | 0.0 | 0.0 | 0.0 | 0.9
  Acute coronary syndrome | 0.4 | 0.0 | 0.0 | 0.0
  Acute myocardial infarction | 0.0 | 0.0 | 0.4 | 0.0
  Angina unstable | 0.4 | 0.0 | 0.0 | 0.0
  Myocardial infarction | 0.4 | 0.0 | 0.0 | 0.0
  Ventricular extrasystoles | 0.4 | 0.4 | 0.0 | 0.4
  Alanine aminotransferase increased | 0.4 | 0.0 | 0.0 | 0.0
  Aspartate aminotransferase increased | 0.0 | 0.0 | 0.0 | 0.4
  Blood creatine phosphokinase increased | 0.0 | 0.0 | 0.0 | 0.4
  Electrocardiogram ST segment depression | 0.0 | 0.4 | 0.0 | 0.0
  Electrocardiogram T wave inversion | 0.4 | 0.0 | 0.0 | 0.0
  Gamma-glutamyltransferase increased | 0.4 | 0.0 | 0.0 | 0.0

61. Secondary Outcome: Absolute Plasma Concentrations
Description: Absolute plasma concentrations of Olodaterol. Values presented are across visits and summarised into geometric means.
Time Frame: within 2 hours before first study drug administration and 10 minutes post-dose at week 6, 12 and 18
Population: Pharmacokinetic set includes all patients in the treated set who had at least one valid olodaterol plasma concentration measurement after initial administration of study drug. This set is restricted to patients in either the Olodaterol 5 μg or 10 μg dose group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 0 | 182 | 216 | 0
pg/mL |  | 3.920 (50.510) | 6.977 (68.643) |

62. Primary Outcome: Mahler Transitional Dyspnea Index Focal Score at 24 Weeks for Combined Analysis
Description: This outcome measure describes the combined analysis of the trials NCT00793624 and NCT00796653. Mahler Transitional Dyspnea Index (TDI) focal score measures 3 components of dyspnea that evoke dyspnea in daily living: Functional Impairment, Magnitude of Task, and Magnitude of Effort. The TDI measures the change from the baseline assessment ranging from -9 (most deterioration) to +9 (most improvement).
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 413 | 433 | 427 | 417
score on a scale | 1.471 (0.155) | 1.980 (0.175) | 1.996 (0.170) | 1.827 (0.168)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Olo 5mcg minus placebo; Test type: Superiority or Other; p = 0.0270, pattern mixture model; See Hogan, et. al. Hogan JW, Roy J, Korkontzelou C Tutorial in biostatistics:handling drop-out in longitudinal studies. Stat Med 23,1455-1497(2004); Mean Difference (Final Values) = 0.509, 95% CI 2-sided [0.058 to 0.960], Standard Error of Mean 0.230 — Based on a pattern mixture model with four patterns based on time of dropout (i.e., day of last observed data) 1) day 43 or day 85, 2) day 127 or day 169, 3) day 225 or day 281, 4) day 337
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Olo 10 mcg minus placebo; Test type: Superiority or Other; p = 0.0203, pattern mixture model; [statistical method as in outcome 62, analysis 1]; Mean Difference (Net) = 0.525, 95% CI 2-sided [0.082 to 0.967], Standard Error of Mean 0.226 — [estimate comment as in outcome 62, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Form 12mcg minus placebo; Test type: Superiority or Other; p = 0.1166, pattern mixture model; [statistical method as in outcome 62, analysis 1]; Mean Difference (Net) = 0.355, 95% CI 2-sided [-0.088 to 0.799], Standard Error of Mean 0.226 — [estimate comment as in outcome 62, analysis 1]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Form 12 mcg
Serious Adverse Events (participants affected / at risk) | 48/235 | 34/232 | 41/234 | 36/233
Other Adverse Events (participants affected / at risk) | 100/235 | 103/232 | 101/234 | 105/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=235) | Olodaterol (Olo) 5 mcg qd (N=232) | Olodaterol (Olo) 10 mcg qd (N=234) | Form 12 mcg (N=233)
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis pharyngeal (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 7 | 4
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 18 | 14 | 17 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Mastoidectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 1
Venous occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=235) | Olodaterol (Olo) 5 mcg qd (N=232) | Olodaterol (Olo) 10 mcg qd (N=234) | Form 12 mcg (N=233)
Pyrexia (General disorders) | 7 | 6 | 12 | 9
Bronchitis (Infections and infestations) | 7 | 13 | 10 | 8
Nasopharyngitis (Infections and infestations) | 22 | 36 | 28 | 23
Upper respiratory tract infection (Infections and infestations) | 18 | 14 | 15 | 21
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 51 | 40 | 48 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 6 | 12 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 3 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication